CLINICAL TRIAL: NCT01826032
Title: Obstructive Sleep Apneas in Elderly:Neuroimaging Changes and Neurocognitive Function Before and After Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Jose M. Montserrat, MD, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OSA-E1
Record Dates: First submitted 2013-03-22; First posted 2013-04-08 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPAP (Experimental): Patients with CPAP treatment. Titration will be performed by polysomnography or automatic CPAP to determine the optimal treatment pressure.
  This group will also be instructed in hygienic-dietary measures and sleep hygiene counselling.
  Interventions: Device: CPAP; Other: Standard care for OSA
- Standard care for OSA (Active Comparator): Sleep hygiene ( regular sleep schedule, avoid sedative drugs, alcohol and tobacco, physical exercise) and dietary counselling
  Interventions: Other: Standard care for OSA

INTERVENTIONS:
Device: CPAP — CPAP treatment every night plus standard care for OSA: lifestyle, and sleep hygiene counselling
  Arms: CPAP
Other: Standard care for OSA — sleep higiene and dietary counseling

SUMMARY:
In the near future more than 20% of the European population will be over 65 years old and the prevalence of obstructive sleep apnea (OSA) in this aged population is known to be higher than 50%. OSA is a risk factor for cognitive dysfunction in middle-aged subjects, but the relationship between cognitive impairment and sleep breathing disorders (SBD) in the elderly has scarcely been observed.

The aim of this study is to investigate cognitive performance in elderly OSA patients, the corresponding brain morphology changes and biological markers and their reversibility with continuous positive airway pressure (CPAP) treatment.

DETAILED DESCRIPTION:
Patients: We will include consecutive patients with a diagnosis of severe OSA (AHI> 30) without significant comorbidities or excessive daytime sleepiness (Epworth ≤ 12). Patients will be randomized to CPAP treatment or conservative treatment.

Methodology: We will assess at baseline and after 3 months of treatment:

1. Neuroimaging by MRI
2. Neurocognitive function with an extensive neuropsychological battery assessing principally memory, attention and executive functions (Trail-making test A and B, Rey Auditory Verbal Learning Test, Digit span, Digit symbol),
3. Biological markers of inflammation and endothelial dysfunction.

Patients included in the study will be monitored and followed for three months. They will be examined at the time of inclusion, after two and six weeks and at the end (12 weeks) for clinical monitoring and the evaluation of adaptation to treatment and compliance.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 65 years old.
2. Patients diagnosed with OSA with an apnea-hypopnea index per hour >30.
3. Patients with an Epworth Sleep Scale score ≤ 12 (without excessive daytime sleepiness).
4. Signed written informed consent.

Exclusion Criteria:

1. Patients with severe chronic diseases: cardiovascular or pulmonary, neurological (stroke, epilepsy, head injury...) or psychiatric.
2. Any current significant systemic illness or unstable medical condition that could lead to difficulty in complying with the protocol or may, in the opinion of the investigator, compromise the conclusions.
3. Mini Mental State Exam (MMSE) <24.
4. Any MRI exclusions - presence of aneurysm clips, pacemakers, mechanic heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body.
5. Previous CPAP treatment.
6. Psycho-physical inability to complete questionnaires. Inadequate visual and auditory acuity will be excluded.
7. Presence of any previously diagnosed sleep disorders: narcolepsy, insomnia, chronic sleep deprivation, REM behavior disorder and restless leg syndrome.
8. Patients with > 50% of central apneas or the presence of Cheyne-Stokes Respiration.
9. History of alcohol abuse or dependence.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Structural and functional brain changes | at baseline and after 3 months of treatment

SECONDARY OUTCOMES:
Assessment of the changing of the neuropsychological tests. | at baseline and after 3 months of treatment
OSA symptoms (daytime sleepiness and everyday function) and quality of life | at baseline and after 3 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Josep M Montserrat, MD, Principal Investigator — Spanish Research Center for Respiratory Diseases
Locations (1):
- Hospital Clinic Barcelona, Barcelona, Catalonia, Spain

REFERENCES:
- [Derived] Dalmases M, Sole-Padulles C, Torres M, Embid C, Nunez MD, Martinez-Garcia MA, Farre R, Bargallo N, Bartres-Faz D, Montserrat JM. Effect of CPAP on Cognition, Brain Function, and Structure Among Elderly Patients With OSA: A Randomized Pilot Study. Chest. 2015 Nov;148(5):1214-1223. doi: 10.1378/chest.15-0171. PMID 26065720